CLINICAL TRIAL: NCT01583868
Title: A Study to Evaluate the Product Feasibility of Two New Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 755E
Record Dates: First submitted 2012-04-23; First posted 2012-04-24 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- B&L RD2135-01 lens C (Experimental): Investigational Silicone hydrogel soft contact lens
  Interventions: Device: B&L RD2135-01 lens C
- B&L RD2135-01 lens D (Experimental): Investigational Silicone hydrogel soft contact lens
  Interventions: Device: B&L RD2135-01 lens D
- PureVision2 (Active Comparator): Bausch & Lomb High definition soft contact lenses
  Interventions: Device: PureVision2
- Ciba Vision Air Optix Aqua (Active Comparator): Ciba Vision Air Optix Aqua soft contact lens
  Interventions: Device: Air Optix Aqua

INTERVENTIONS:
Device: B&L RD2135-01 lens C — Lenses will be worn on a daily wear basis for 1 week. Lens care solution and lens cases will be provided for daily rinsing, cleaning, disinfecting, and storing the lenses. Rewetting drops will be provided for use as needed during the study.
  Arms: B&L RD2135-01 lens C
Device: B&L RD2135-01 lens D — Lenses will be worn on a daily wear basis for 1 week. Lens care solution and lens cases will be provided for daily rinsing, cleaning, disinfecting, and storing the lenses. Rewetting drops will be provided for use as needed during the study.
  Arms: B&L RD2135-01 lens D
Device: PureVision2 — Lenses will be worn on a daily wear basis for 1 week. Lens care solution and lens cases will be provided for daily rinsing, cleaning, disinfecting, and storing the lenses. Rewetting drops will be provided for use as needed during the study.
  Arms: PureVision2
Device: Air Optix Aqua — Lenses will be worn on a daily wear basis for 1 week. Lens care solution and lens cases will be provided for daily rinsing, cleaning, disinfecting, and storing the lenses. Rewetting drops will be provided for use as needed during the study.
  Arms: Ciba Vision Air Optix Aqua

SUMMARY:
The objective of this study is to determine the clinical feasibility and to evaluate the product performance of two RD2135-01 investigational soft contact lenses (Test 1 and Test 2) developed by Bausch + Lomb. The Test lenses will be compared to both Bausch + Lomb PureVision®2 HD (high definition) soft contact lenses and Ciba Vision Air Optix Aqua soft contact lenses when used among currently adapted soft contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
* Be adapted wearers of soft contact lenses, wear a lens in each eye, and each lens must be of the same manufacture and brand.
* Be correctable through spherocylindrical refraction to 32 letters (0.3 logMAR) or better (distance, high contrast) in each eye.
* Be myopic and require lens correction from -0.50 diopters (D) to -6.00 D in each eye.
* Must agree to wear the study lenses on a daily wear basis for the duration of the study.
* Must be willing to use a lens care system on a regular basis.
* If the subject requires a Washout Period, the subject must be willing to discontinue contact lens wear and be willing to wear either spectacles or no lenses during this Washout Period.

Exclusion Criteria:

* Not correctable to 32 letters (0.3 logMAR) in each eye with soft spherical contact lenses.
* Have an active ocular disease, any corneal infiltrative response or are using any ocular medications.
* Have worn gas permeable (GP) contact lenses within last 30 days or PMMA lenses within last 3 months.
* Any scar or neovascularization within the central 4mm of the cornea.
* Any Grade 2 or greater finding during the slit lamp examination, Subjects with corneal infiltrates, of ANY GRADE, are not eligible.
* Any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Anisometropia (spherical equivalent) of greater than 2.00 D.
* Any systemic disease affecting ocular health.
* Using any systemic or topical medications that will affect ocular physiology or lens performance.
* Aphakic.
* Amblyopic.
* Allergic to any component in the study products.
* Have had any corneal surgery (ie, refractive surgery).
* Currently wear monovision correction, multifocal, or toric contact lenses.
* Ocular astigmatism greater than 1.00 D in either eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly J Barna, CCRA, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, bilateral, study, with a crossover at one week and a second crossover at two weeks. A total of 216 subjects (432 eyes) were enrolled in this study. Participants were randomized to receive either, the Test Lens C, Test Lens D and PureVision2 lenses, or the Test Lens C, Test Lens D and Air Optix Aqua lenses.
Groups:
- B&L RD2135-01 Lens C Then B&L RD2135-01 Lens D Then PureVision: B&L RD2135-01 Lens C for one week then B&L RD2135-01 Lens D for one week then PureVision2 for one week
- B&L RD2135-01 Lens C Then B&L RD2135-01 Lens D Then Ciba Vis: B&L RD2135-01 Lens C for one week then B&L RD2135-01 Lens D for one week then Ciba Vision for one week
Period: Overall Study
Arm/Group | B&L RD2135-01 Lens C Then B&L RD2135-01 Lens D Then PureVision | B&L RD2135-01 Lens C Then B&L RD2135-01 Lens D Then Ciba Vis
Started | 108 | 108
Completed | 104 | 104
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: Demography was collected for 210 eligible, dispensed participants. Participants received multiple treatment groups in this cross-over study. Two participants did not have demography information.
Groups:
- Total: Total of all reporting groups
Arm/Group | B&L RD2135-01 Lens C Then B&L RD2135-01 Lens D Then PureVision | B&L RD2135-01 Lens C Then B&L RD2135-01 Lens D Then Ciba Vis | Total
Number analyzed (Participants) | 105 | 105 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (8.55) | 31.8 (8.68) | 31.5 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 71 | 143
  Male | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Visual acuity was assessed by distance high contrast logarithm of the minimum angle of resolution (logMAR).
Time Frame: At 1 week follow up
Population: There were 212 eligible, dispensed participants (424 eyes). Participants/eyes received multiple treatment groups in this cross-over study. All eyes received investigational lens C and investigation lens D. Half of the eyes received PureVision2 and half of the eyes received Ciba Vision Air Optix Aqua.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | B&L RD2135-01 Lens C | B&L RD2135-01 Lens D | PureVision2 | Ciba Vision Air Optix Aqua
Number analyzed (Participants) | 212 | 212 | 106 | 106
Number analyzed (eyes) | 424 | 424 | 212 | 212
logMAR | -0.089 (0.078) | -0.087 (0.079) | -0.086 (0.077) | -0.086 (0.082)

2. Secondary Outcome: Symptoms and Complaints
Description: Symptoms/complaints were assessed on a scale from 0 to 100, with 0 denoting unfavorable symptoms/complaints. Symptoms/complaints were recorded for each eye based on the participant's experience with their study lenses worn for that respective treatment period. Symptoms/complaints parameters included the following: Burning/stinging upon insertion, Comfort upon insertion, Overall comfort, Comfort at end of day, Ease of handling/insertion, Ease of handling/removal, Dryness, Itchiness, Redness, Vision upon insertion, Vision, Vision in low light, Lens cleanness upon insertion, Lens cleanness upon removal, Lens cleanness, Dryness at end of day, and Overall impression.
Time Frame: At 1 Week follow up
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | B&L RD2135-01 Lens C | B&L RD2135-01 Lens D | PureVision2 | Ciba Vision Air Optix Aqua
Number analyzed (Participants) | 212 | 212 | 106 | 106
Number analyzed (eyes) | 424 | 424 | 212 | 212
score on a scale
  Burning/stinging upon insertion | 91.3 (13.1) | 91.3 (12.4) | 83.1 (21.4) | 92.6 (9.9)
  Comfort upon insertion | 89.6 (14.5) | 88.2 (15.6) | 78.7 (15.6) | 89.6 (12.0)
  Overall comfort | 88.0 (14.6) | 85.7 (16.9) | 78.4 (20.4) | 86.6 (15.8)
  Comfort at end of day | 81.2 (18.9) | 79.3 (20.2) | 72.0 (22.9) | 79.7 (19.7)
  Ease of handling/insertion | 89.5 (16.6) | 88.6 (17.3) | 85.0 (20.4) | 89.0 (15.3)
  Ease of handling/removal | 91.1 (14.3) | 91.0 (13.6) | 89.4 (15.6) | 89.4 (15.5)
  Dryness | 84.4 (16.1) | 81.9 (18.1) | 77.0 (21.6) | 84.4 (17.3)
  Itchiness | 90.6 (12.9) | 89.6 (15.9) | 87.4 (17.0) | 88.5 (17.3)
  Redness | 92.4 (11.7) | 91.6 (13.1) | 90.6 (14.0) | 91.2 (12.5)
  Vision upon insertion | 93.4 (9.6) | 91.5 (13.3) | 87.0 (17.5) | 93.1 (9.6)
  Vision | 92.3 (11.4) | 91.9 (13.1) | 88.1 (14.6) | 93.5 (10.3)
  Vision in low light | 91.0 (11.9) | 89.9 (13.4) | 87.3 (13.8) | 91.4 (12.5)
  Lens cleanness upon insertion | 93.1 (10.9) | 92.8 (11.4) | 89.7 (14.6) | 94.4 (7.7)
  Lens cleannes upon removal | 89.9 (12.2) | 89.3 (12.9) | 86.3 (17.2) | 90.9 (9.7)
  Lens cleanness | 91.8 (10.6) | 91.2 (11.7) | 86.6 (17.0) | 92.5 (9.1)
  Dryness at end of day | 82.4 (17.7) | 80.3 (19.3) | 75.5 (21.7) | 82.4 (17.3)
  Overall impression | 84.5 (17.0) | 82.2 (19.0) | 73.7 (24.6) | 83.9 (18.3)

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: Adverse events (AEs) were not coded. Therefore, source vocabulary is not applicable. Safety data were collected for 212 eligible, dispensed participants. Participants received multiple treatment groups in this cross-over study.
Groups:
- B&L RD2135-01 Lens C: B&L RD2135-01 Lens C
- B&L RD2135-01 Lens D: B&L RD2135-01 Lens D
- PureVision2: PureVision2
- Ciba Vision Air Optix Aqua: Ciba Vision Air Optix Aqua
Arm/Group | B&L RD2135-01 Lens C | B&L RD2135-01 Lens D | PureVision2 | Ciba Vision Air Optix Aqua
Serious Adverse Events (participants affected / at risk) | 0/212 | 0/212 | 0/106 | 0/106
Other Adverse Events (participants affected / at risk) | 0/212 | 0/212 | 0/106 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.